CLINICAL TRIAL: NCT01728389
Title: Efficacy and Safety of Direct Intrabone Transplantation of Peripheral Blood Haematopoietic Stem Cells Form HLA-matched Sibling Donors in Patients With Myeloid and Lymphoid Malignancies.
Brief Title: Intrabone Transplantation of Allogenic Peripheral Blood Stem Cells in Patients With Myeloid and Lymphoid Malignancies.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBT-COI-01
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Leukemia; Lymphoma
Keywords: allogenic stem cell transplantation; peripheral blood stem cells; intrabone; intra-bone; leukemia; lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intrabone transplantation (Experimental): Direct intrabone transplantation procedure of peripheral blood haematopoietic stem cells form HLA-matched sibling donors in patients with myeloid and lymphoid malignancies.
  Interventions: Procedure: Intrabone transplantation

INTERVENTIONS:
Procedure: Intrabone transplantation — Direct intrabone transplantation procedure of peripheral blood haematopoietic stem cells form HLA-matched sibling donors in patients with myeloid and lymphoid malignancies.

SUMMARY:
The purpose of the study is to evaluate efficacy and safety of direct intrabone transplantation procedure of peripheral blood haematopoietic stem cells form HLA-matched sibling donors in patients with myeloid and lymphoid malignancies.

DETAILED DESCRIPTION:
Allogenic haematopoietic stem cell transplantation is an established treatment option for haematologic malignancies, especially leukaemias and lymphomas, providing curative potential. The optimal donor is HLA-matched sibling and G-CSF stimulated peripheral blood is nowadays the most common source of stem cells. Routinely used route of stem cell transplantation is intravenous infusion via central venous catheter. Based on the animal studies, only 10-15% of intravenously transplanted stem cells migrate to haematopoietic sites while the rest is lost in other organs. Results of studies of direct intrabone allogenic cord-blood cells transplantation in humans confirm that this route of transplantation is associated with less probability of graft failure and moreover may reduce risk of graft-versus-host disease and malignancy relapse. For those purposes in the current study we investigate intrabone route of allogenic peripheral blood stem cell transplantation. Our intention is to achieve fast engraftment and minimize risk of relapse and graft graft-versus-host disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Diagnosis of leukaemia or lymphoma
* Indication for allogenic stem cell transplantation according to European Group for Blood and Marrow Transplantation guidelines
* HLA-matched sibling donor qualified for peripheral blood stem cell donation
* Performance status WHO 0-1
* Written informed consent

Exclusion Criteria:

* Organ dysfunction: elevated ALT, AST, bilirubin, AF; creatinine >1.5 upper normal limit; LVEF <45%
* Active infection
* Unstable diabetes
* Psychiatric diseases
* Obesity or anatomical obstacle for direct intrabone transplantation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Neutrophil engraftment (ANC > 0,5 G/l) | 28 days

SECONDARY OUTCOMES:
Lineage chimerism of peripheral blood T-cell lymphocytes | 1 year
Platelet engraftment (Plt > 20 G/l) | 28 days
Adverse reactions related with intrabone transplantation procedure | 28 days

OTHER OUTCOMES:
Relapse incidence | 1 year
Overall survival | 1 year
Disease-free survival | 1 year
Graft-versus-host disease incidence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Czerw, MD, Principal Investigator — Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland
Locations (1):
- MSC Memorial CAncer Center and Institute of Oncology, Gliwice, Poland

REFERENCES:
- [Background] Frassoni F, Gualandi F, Podesta M, Raiola AM, Ibatici A, Piaggio G, Sessarego M, Sessarego N, Gobbi M, Sacchi N, Labopin M, Bacigalupo A. Direct intrabone transplant of unrelated cord-blood cells in acute leukaemia: a phase I/II study. Lancet Oncol. 2008 Sep;9(9):831-9. doi: 10.1016/S1470-2045(08)70180-3. Epub 2008 Aug 8. PMID 18693069
- [Background] Okada M, Yoshihara S, Taniguchi K, Kaida K, Ikegame K, Kato R, Tamaki H, Inoue T, Soma T, Kai S, Kato S, Ogawa H. Intrabone marrow transplantation of unwashed cord blood using reduced-intensity conditioning treatment: a phase I study. Biol Blood Marrow Transplant. 2012 Apr;18(4):633-9. doi: 10.1016/j.bbmt.2011.08.010. Epub 2011 Aug 23. PMID 21867667
- [Background] Massollo M, Podesta M, Marini C, Morbelli S, Cassanelli C, Pinto V, Ubezio G, Curti G, Uccelli A, Frassoni F, Sambuceti G. Contact with the bone marrow microenvironment readdresses the fate of transplanted hematopoietic stem cells. Exp Hematol. 2010 Oct;38(10):968-77. doi: 10.1016/j.exphem.2010.06.003. Epub 2010 Jun 13. PMID 20550953